CLINICAL TRIAL: NCT04166474
Title: Drug Interactions Between Dolutegravir and Escalating Doses of Rifampicin
Acronym: DoRIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helen Reynolds (Other)
Collaborators: Infectious Disease Institute, Kampala, Uganda (Other); Desmond Tutu HIV Centre (Other)
Responsible Party: Sponsor-Investigator, Helen Reynolds, Programme manager, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UoL001452
Record Dates: First submitted 2019-11-01; First posted 2019-11-18 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hiv; Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dolutegravir (Experimental)
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Dosed at 50 mg bd on 3 separate occasions with low, medium and high doses of rifampicin. Dosed at 50 mg od without rifampicin.

SUMMARY:
This is a drug interaction study in HIV negative, TB-monoinfected participants coming to the end of continuation phase of TB therapy, to study the pharmacokinetic changes to dolutegravir when administered with standard, medium and high dose rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent prior to participation
* Willing and able to comply with all study requirements
* Receiving standard doses of RIF and INH
* HIV antibody negative
* Male or non-pregnant, non-breastfeeding female
* Study participation will not extend length of ATT by more than 4 weeks

Exclusion Criteria:

* < 18 years
* Body weight < 50 kg
* eGFR < 60 mL/min
* Abnormal LFTs including ALT > 2.5 ULN
* HIV antibody positive
* Non-standard TB regimen (containing RHZE)
* Women of childbearing age unless using effective contraception
* Family history of sudden cardiac death
* Prior history of cardiac disease that precludes the use of low dose digoxin
* Medical or psychiatric condition that might affect participation in the study based on investigator judgement
* Regular consumption of grapefruit or grapefruit juice
* ECG abnormalities that preclude the use of low dose digoxin (intermittent complete heart block, second degree AV block, supraventricular arrhythmia associated with conducting pathways, ventricular tachycardia or fibrillation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Change in pharmacokinetic parameter Cmin of dolutegravir | Day 14, Day 28, Day 42, 5 weeks post anti-tuberculosis treatment
  Change in dolutegravir Cmin when dosed with standard, medium, high dose rifampicin

SECONDARY OUTCOMES:
Change in pharmacokinetic parameter AUC of dolutegravir | Day 14, Day 28, Day 42, 5 weeks post anti-tuberculosis treatment
  Change in dolutegravir AUC when dosed with standard, medium, high dose rifampicin
Change in pharmacokinetic parameter Cmax of dolutegravir | Day 14, Day 28, Day 42, 5 weeks post anti-tuberculosis treatment
  Change in dolutegravir Cmax when dosed with standard, medium, high dose rifampicin
Number of participants with Grade 3 and above adverse events as assessed by DAIDS (corrected v2.1 July 2017) | From first dose of dolutegravir until study completion approximately 2 years
  Number of participants with Grade 3 and above adverse events as assessed by DAIDS (corrected v2.1 July 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Saye Khoo, Principal Investigator — University of Liverpool
Locations (2):
- Desmond Tutu Health Foundation, Cape Town, South Africa
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No